CLINICAL TRIAL: NCT00281619
Title: Development of Population Pharmacokinetic-Pharmacodynamic (PK-PD) Models of Mycophenolic Acid for Bayesian Dose Individualization in Pediatric Kidney Transplant Patients
Brief Title: PK-PD Study of Mycophenolic Acid (CellCept) in Pediatric Kidney Transplant Patients
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: CEL420 MPA (PK-PD); CEL420
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Kidney Transplant
Keywords: Pediatric Kidney Transplant; Kidney Transplant; CellCept; Mycophenolate mofetil; Mycophenolic Acid; MPA
MeSH Terms: interventions — Mycophenolic Acid; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mycophenolic Acid (CellCept): purpose of this study is to determine how fast children, who have had a recent kidney transplant, absorb, breakdown and eliminate mycophenolic acid (CellCept) following their prescribed dose
  Interventions: Drug: CellCept (mycophenolate mofetil); Behavioral: Dietary Monitoring; Behavioral: Drug Diary; Procedure: Blood Sampling

INTERVENTIONS:
Drug: CellCept (mycophenolate mofetil)
Behavioral: Dietary Monitoring
Behavioral: Drug Diary
Procedure: Blood Sampling

SUMMARY:
The purpose of this study is to determine how fast children, who have had a recent kidney transplant, absorb, breakdown and eliminate mycophenolic acid (CellCept) following their prescribed dose. The results may lead to better dosing based on individual needs.

DETAILED DESCRIPTION:
This is an open-label, inpatient-outpatient population pharmacokinetic-pharmacodynamic (PK-PD) study of mycophenolic acid (MPA) in pediatric subjects (age 2-17 years) who have had a recent kidney transplant, as well as during the stable renal transplant period when on a stable oral regimen of MPA. The primary objective of this study is to develop population pharmacokinetic-pharmacodynamic (PK-PD) models for mycophenolic acid (MPA) and mycophenolic acid glucuronide (MPAG) in order to improve individualized pediatric dosing. Subjects will have been receiving CellCept as part of their clinical standard of care. It is anticipated that the clinical portion of the study for each patient will be approximately six months post renal transplant with four study days: a screening visit pre-transplant, two 10-hour inpatient days at 2-3 and 6-9 days post-transplant, and one (up to 10 hour) outpatient visit at 3-6 months post-transplant. Pharmacokinetic and pharmacodynamic measurements will be conducted at various time points (up to 9 hours post dose) on study days 2, 3, and 4. Safety data to be collected will include physical examinations, measurement of vital signs, and laboratory assessments, as well as data on adverse events and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects and non-pregnant female subjects aged 2 to 17 years who are about to receive a kidney transplant and will be on post transplant MMF containing immunosuppressive therapy. Subjects may be enrolled up to their 18th year.
* Minimum weight of 11 kg.
* A signed and dated IRB approved parental / guardian informed consent form and an IRB-approved child assent form if applicable.
* A high probability for compliance with and completion of the study.
* For post-transplant study period: Subjects with stable kidney allografts who are at least 3 months post-transplant and who have received the same regimen of MMF (with cyclosporine or tacrolimus) for at least 30 days before the study visit (3-6 months post-transplant).
* May have clinically important abnormalities on clinical and /or laboratory evaluations only as these abnormalities relate to an underlying condition as determined by the principal investigator.
* Other variations from established normal ranges may be acceptable if they are not clinically significant in the opinion of the investigators.

Exclusion Criteria:

* Any medical condition (active or chronic) or prior surgery that may interfere with the pharmacokinetic behavior of MMF (absorption, distribution and elimination) as determined by the PI.
* Active systemic infection.
* History of substance abuse.
* Signs or symptoms of active hepatitis (a history of hepatitis B or C virus infection is permitted).
* Known history of or suspected infection with human immunodeficiency virus (HIV).

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Male subjects and non-pregnant female subjects aged 2-17 years who are about to receive a kidney transplant and will be on post transplant MMF containing immunosuppressive therapy, per clinical care.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2006-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
The following outcome measures will be performed at study visit 2 (2-3 days post-transplant), study visit 3 (6-9 days post-transplant), and study visit 4 (3-6 months post-transplant): | 6 months
Drug Measurement of MPA and MPA-G | 6 months
IMPDH Assay | 6 months
Mitogenesis Assays and | 6 months
Determination of CD25 Expression. | 6 months

SECONDARY OUTCOMES:
Concomitant medications and MPA (CellCept) drug diary (study visits 1-4) | 6 months
Physical Exam (study visits 1-4) | 6 months
Safety Laboratory tests (study visits 1-4) | 6 months
Dietary Monitoring (study visits 2,3 & 4) | 6 months
Adverse Event Reporting (study visits 1-4). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander A. Vinks, PharmD., PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States